CLINICAL TRIAL: NCT00745797
Title: Prophylactic Cranial Irradiation (PCI) Versus no PCI in Non Small Cell Lung Cancer After a Response to Chemotherapy：A Multi-center Randomized Phase ⅢTrial
Brief Title: Prophylactic Cranial Irradiation (PCI) Versus no PCI in Non Small Cell Lung Cancer After a Response to Chemotherapy
Acronym: PCI
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: this trial enroll extremely slow and No funding support
Sponsor: Yi-Long Wu (Other)
Responsible Party: Sponsor-Investigator, Yi-Long Wu, Professor, director, Chinese Society of Lung Cancer
Organization: Chinese Society of Lung Cancer (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CSLC0801
Record Dates: First submitted 2008-09-02; First posted 2008-09-03 (Estimated); Last update posted 2017-03-06 (Actual); Status verified 2017-03

CONDITIONS: Brain Metastases
Keywords: nonsmall cell lung cancer; brain metastasis; prophylactic cranial irradiation
MeSH Terms: conditions — Brain Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prophylactic WBRT (Experimental): Take the whole brain radiotherapy radiotherapy
  Interventions: Radiation: Radiotherapy
- Observer Group (No Intervention): The first 14 days after randomization and patient follow-up after 1 month to complete the FACT-L questionnaire and the MMSE scale.

INTERVENTIONS:
Radiation: Radiotherapy — blood transfusions, platelet transfusions, antibiotics, antipyretic analgesics and anesthetics
  Other Names: Radiotherapy,Dehydration drugs, elevated white blood drugs,
  Arms: Prophylactic WBRT

SUMMARY:
1. Patients with confirmed advanced NSCLC and any response to 3-6 cycles of chemotherapy, were randomized to receive PCI (30 Gy/10fr) or no PCI.
2. The primary endpoint was the cumulative incidence of symptomatic brain metastases (BM) .
3. The study was sized to detect a hazard ratio of 0.37 with 80% power and 2-sided 5% significance (60 events, 206 patients).

DETAILED DESCRIPTION:
1. Prophylactic cranial irradiation (PCI) significantly reduces the risk of brain metastases (BM) and improves survival in patients with extensive disease small cell lung cancer after a response to chemotherapy .
2. PCI has also demonstrated to reduce or delay the incidence of CNS failure in non small cell lung cancer patients after primary therapy.
3. But its impact on overall and disease free survival is uncertain.

ELIGIBILITY:
Inclusion Criteria:

1. Patients were required to have histologically or cytologically documented NSCLC and no brain metastasis documented by magnetic resonance imaging (MRI)within 21 days after confirmed response (RR+SD) to chemotherapy
2. No previous history of radiotherapy and surgery of brain
3. Agree to radiotherapy
4. age > 18 and <75 years
5. ECOG performance status 1 or less
6. Good renal and hepatic and haematological (absolute neutrophils count 15 x1O9/L and platelet count 90 x 109/L,HB>=80g /DL) functions
7. Have provided informed consent

Exclusion Criteria:

1. Seizure cannot be controled by the drugs
2. Combined with other disease of the brain such as tumour or infarction
3. Hypersensitivity to MR enhancer

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2008-04; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is the cumulative incidence of symptomatic brain metastases (BM) . | 2.5years

SECONDARY OUTCOMES:
1year survival,overall survival,incidence rate of radioactive brain injured | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: WU YI LONG, MD, Principal Investigator — Chinese Society of Lung Cancer
Locations (1):
- Lung Cancer Research Institute & Cancer Center of Guangdong Provincial People's Hospital, Guangzhou, Guangdong, China